CLINICAL TRIAL: NCT01012167
Title: Oxytocin or Galantamine vs. Placebo for the Treatment of Negative Symptoms and Cognitive Impairments in Schizophrenia
Brief Title: Oxytocin or Galantamine Versus Placebo for the Treatment of Negative Symptoms and Cognitive Impairments in Schizophrenia
Acronym: CIDAR-3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Robert Buchanan, Chief, Maryland Psychiatric Research Center, Outpatient Research Program, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HP-00044324; 1P50MH082999-01 (NIH)
Record Dates: First submitted 2009-04-28; First posted 2009-11-11 (Estimated); Results first posted 2017-06-02 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2022-01

CONDITIONS: Schizophrenia
Keywords: Schizophrenia, oxytocin, galantamine
MeSH Terms: conditions — Schizophrenia | interventions — Oxytocin; Galantamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1: galantamine/placebo-oxytocin (Active Comparator): Subjects randomized to galantamine will receive galantamine and placebo-oxytocin
  Interventions: Drug: Galantamine; Other: Placebo-Oxytocin
- 2: oxytocin/placebo-galantamine (Active Comparator): Subjects randomized to oxytocin will receive oxytocin and placebo-galantamine
  Interventions: Drug: Oxytocin; Other: Placebo-Galantamine
- 3: placebo-galantamine /placebo-oxytocin (Placebo Comparator): Subjects randomized to placebo will receive placebo-galantamine and placebo-oxytocin
  Interventions: Other: Placebo-Oxytocin; Other: Placebo-Galantamine

INTERVENTIONS:
Drug: Oxytocin — Oxytocin: 24 IU in the morning and 24 IU in the evening given by nasal spray with a total of 6 puffs of the spray, 3 in each nostril at each administration
  Arms: 2: oxytocin/placebo-galantamine
Drug: Galantamine — Galantamine: 4 mg twice a day for 1 week, then 8 mg twice a day for 1 week, then 12 mg twice a day for 4 weeks
  Arms: 1: galantamine/placebo-oxytocin
Other: Placebo-Oxytocin — Saline nasal spray with a total of 6 puffs of the spray, 3 in each nostril at each administration
  Arms: 1: galantamine/placebo-oxytocin; 3: placebo-galantamine /placebo-oxytocin
Other: Placebo-Galantamine — Placebo tablets twice a day for 6 weeks
  Arms: 2: oxytocin/placebo-galantamine; 3: placebo-galantamine /placebo-oxytocin

SUMMARY:
The project is designed to address the following two primary aims:

1. To determine whether adjunctive oxytocin is superior to placebo for the treatment of persistent negative symptoms, as measured by the SANS total score, in people with schizophrenia.
2. To determine whether adjunctive Galantamine is superior to placebo for the treatment of cognitive impairments, as measured by improvement on a composite neurocognitive score in people with schizophrenia.

The investigators will also address the following secondary aims:

1. To determine whether people with schizophrenia treated with adjunctive oxytocin, compared to placebo, will show greater improvement on markers of negative symptom liability including: social affiliation, facial affect recognition, olfactory discrimination, initiation of smooth pursuit and latency of internally-driven saccades.
2. To determine whether people with schizophrenia treated with adjunctive Galantamine, compared to placebo, will show greater improvement on markers of cognitive impairment liability including: predictive pursuit, P50 sensory gating and visual-spatial working memory.

The investigators will address the following exploratory aims:

1. To determine whether changes in markers of negative symptom liability are correlated with changes in SANS total score.
2. To determine whether changes in markers of cognitive impairment liability are correlated with changes in the composite neurocognitive score.
3. To determine the response to oxytocin of all cognition domains assessed by the MATRICS battery, and to determine the response to Galantamine of all cognition domains assessed by the MATRICS, which are not included in the primary neurocognitive outcome score.
4. To determine whether there is a differential response of oxytocin and Galantamine on the SANS total score, composite neurocognitive score, and with the phenotypic measures of negative symptom and cognitive impairment liability.
5. To determine whether oxytocin and Galantamine are associated with:

   * adverse effects on positive or depressive symptoms;
   * adverse effects on motor symptoms;
   * adverse effects on laboratory and EKG measures;
   * increased occurrence of side effects;
   * social interest that is independent of sexual desire.

ELIGIBILITY:
Inclusion Criteria:

* Any race
* Subjects will meet DSM-IV criteria for schizophrenia or schizoaffective disorder
* Judged clinically stable and will not exceed threshold levels of positive, depressive, and/or extrapyramidal symptoms
* The minimum level of negative symptoms will be defined as follows:

  * Scale for the Assessment of Negative Symptoms (SANS) total score (minus the global items, and inappropriate affect, poverty of content of speech and attentional items) 20 or greater; OR
  * SANS alogia global item score 3 or greater
* The maximum level of psychotic, depressive, and extrapyramidal symptoms at the beginning and end of leading in:

  * Brief Psychiatric Rating Scale (BPRS) psychotic factor score (4-items) less or equal to 16
  * BPRS Anxiety/Depression factor score (4-items) less than or equal to 14
  * Simpson-Angus-Scale (SAS) total score (13-items) less than or equal to 10
* Subjects will be required to be on the same antipsychotic(s) for two months and on the same dose for the last month

Exclusion Criteria:

* Participants with an organic brain disorder; mental retardation; or a medical condition, whose pathology or treatment could alter the presentation or treatment of schizophrenia or significantly increase the risk associated with the proposed treatment protocol
* Participants with intermittent alcohol or substance use will not be excluded unless they have met DSM-IV criteria for alcohol or substance abuse (other than nicotine) within the last month.
* Participants may be treated with one or more antipsychotics, except chlorpromazine, thioridazine, or mesoridazine. These latter antipsychotics are excluded because of the concern that their anticholinergic properties may interfere with the accurate assessment of galantamine efficacy.
* Participants may not be treated with anticholinergic medications or have clinically significant extrapyramidal symptoms. Additionally, subjects treated with glycopyrrolate will be accepted.
* Female participants may not be pregnant
* Female subjects may not be taking olanzapine at doses higher than 30 mg . Male subjects may not be taking olanzapine at doses higher than 40 mg.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2010-02; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William T Carpenter, M.D., Principal Investigator — Maryland Psychiatric Research Center
Locations (6):
- United States (6):
  - Baltimore VA Medical Center, Baltimore, Maryland
  - Community Mental Health Centers, Baltimore, Maryland
  - Keypoint Community Mental Health Centers, Baltimore, Maryland
  - Maryland Psychiatric Research Center, Baltimore, Maryland
  - Maryland Psychiatric Research Center, Catonsville, Maryland
  - Keypoint Mental health Center, Dundalk, Maryland

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Consented/Screened for Study-- N=86
  Withdrew prior to randomization (N=28)
  * 2 withdrew consent
  * 26 did not meet inclusion criteria
  Randomized-- N=58
Groups:
- 1: Oxytocin/Placebo-galantamine: Subjects randomized to oxytocin will receive oxytocin and placebo-galantamine
- 2: Galantamine/Placebo-oxytocin: Subjects randomized to galantamine will receive galantamine and placebo-oxytocin
Period: Overall Study
Arm/Group | 1: Oxytocin/Placebo-galantamine | 2: Galantamine/Placebo-oxytocin | 3: Placebo-galantamine /Placebo-oxytocin
Started | 17 | 20 | 21
Withdrawn Prior to Study Drug Exposure | 1 | 0 | 1
Exposed to Study Drug | 16 | 20 | 20
Completed | 15 | 18 | 17
Not Completed | 2 | 2 | 4

BASELINE CHARACTERISTICS:
Population: Number of participants randomized N=58
  Withdrawn prior to exposure to study drug (N=2) Oxytocin N=1 withdrawn due to abnormal EKG Placebo N=1 Participant withdrew consent
  Exposed to study drug N=56
Groups:
- 1: Oxytocin: Oxytocin: 24 IU oxytocin or placebo in a total of 6 puffs (3 puffs per nostril)daily for 6 weeks
- 2: Galantamine: Galantamine or placebo Galantamine: Galantamine will be dispensed as follows: 4 mg bid x 7 days; 8mg bid x 7days, then 12 mg bid for the last 4 weeks.
- 3: Placebo: Placebo: placebo-Galantamine 1 capsules twice a day and placebo-oxytocin 3 puffs in each nostril once a day.
- Total: Total of all reporting groups
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo | Total
Number analyzed (Participants) | 16 | 20 | 20 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 20 | 20 | 56
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.4 (11.2) | 45.8 (12.4) | 42.2 (11.7) | 44.9 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 3 | 11
  Male | 14 | 14 | 17 | 45
Region of Enrollment [Number; unit: participants]
  United States | 16 | 20 | 20 | 56

OUTCOME MEASURES:

1. Primary Outcome: Scale for the Assessment of Negative Symptoms (SANS) Total Score
Description: Mean SANS Total Score by Treatment and Week. SANS total score range = 0-85. Higher scores indicate more severe negative symptoms.
Time Frame: Every other week for 6 weeks
Population: Of the 56 participants exposed to study drug, 3 withdrew before any efficacy data was collected, leaving 53 for whom at least some interim efficacy data was collected. Participants had to complete at least two weeks follow-up to be included in the symptom analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1: Oxytocin/Placebo-galantamine | 2: Galantamine/Placebo-oxytocin | 3: Placebo-galantamine /Placebo-oxytocin
Number analyzed (Participants) | 15 | 19 | 19
units on a scale
  Treatment Week 0 | 33.23 (6.91) | 36.63 (10.09) | 36.63 (10.61)
  Treatment Week 2 | 30.07 (6.93) | 35.22 (10.97) | 35.05 (10.52)
  Treatment Week 4: number analyzed (Participants) | 15 | 18 | 18
  Treatment Week 4 | 31.27 (7.53) | 34.06 (10.26) | 34.22 (9.61)
  Treatment Week 6: number analyzed (Participants) | 15 | 18 | 17
  Treatment Week 6 | 31.40 (6.85) | 33.22 (10.64) | 33.47 (8.47)
  Change from Week 0 at Week 2 | -3.17 (4.20) | -1.41 (3.32) | -1.58 (4.84)
  Change from Week 0 at Week 4: number analyzed (Participants) | 15 | 18 | 18
  Change from Week 0 at Week 4 | -1.97 (4.48) | -1.69 (3.46) | -1.47 (5.64)
  Change from Week 0 at Week 6: number analyzed (Participants) | 15 | 18 | 17
  Change from Week 0 at Week 6 | -1.83 (3.74) | -2.53 (4.34) | -1.00 (4.41)

2. Primary Outcome: Mean Z-Scores for Composite Cognitive Primary Outcome* by Treatment Group and Week
Description: * Composite Cognitive Primary Outcome = mean of z-scores from the Brief Assessment of Cognition in Schizophrenia (BACS) Symbol Digit test, the Hopkins Verbal Learning Test (HVLT), and the Rapid Visual Information Processing test (RVIP). Z-scores for each test were calculated as Z = (individual patient score - pooled baseline mean)/(pooled baseline standard deviation). Higher values of the composite score represent a better outcome.
Time Frame: Treatment Week 0 and Week 6
Population: Five subjects were unable to handle the demands of the Rapid Visual Information Processing (RVIP) test, part of the composite primary outcome measure, and did not provide valid data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1: Oxytocin/Placebo-galantamine | 2: Galantamine/Placebo-oxytocin | 3: Placebo-galantamine /Placebo-oxytocin
Number analyzed (Participants) | 14 | 15 | 16
units on a scale
  Treatment Week 0 | 0.23 (0.92) | -0.22 (0.47) | 0.21 (0.83)
  Treatment Week 6: number analyzed (Participants) | 14 | 15 | 15
  Treatment Week 6 | 0.33 (1) | -0.05 (0.68) | 0.18 (0.69)
  Change: number analyzed (Participants) | 14 | 15 | 15
  Change | 0.1 (0.37) | 0.17 (0.44) | 0.03 (0.41)

3. Secondary Outcome: Scale for the Assessment of Negative Symptoms (SANS) - Avolition
Description: Mean score by treatment and week. Scores range from 0-5, with higher scores indicating a worse outcome.
Time Frame: Every other week for 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1: Oxytocin/Placebo-galantamine | 2: Galantamine/Placebo-oxytocin | 3: Placebo-galantamine /Placebo-oxytocin
Number analyzed (Participants) | 15 | 19 | 19
units on a scale
  Treatment Week 0 | 2.94 (0.90) | 2.91 (0.88) | 2.44 (0.97)
  Treatment Week 2 | 2.78 (0.77) | 2.73 (0.74) | 2.43 (0.93)
  Treatment Week 4: number analyzed (Participants) | 15 | 18 | 18
  Treatment Week 4 | 2.85 (1.04) | 2.74 (.084) | 2.44 (0.94)
  Treatment Week 6: number analyzed (Participants) | 15 | 18 | 17
  Treatment Week 6 | 2.88 (0.89) | 2.74 (0.90) | 2.41 (0.87)
  Change from Week 0 at Week 2 | -0.15 (0.32) | -0.18 (0.43) | -0.01 (0.57)
  Change from Week 0 at Week 4: number analyzed (Participants) | 15 | 18 | 18
  Change from Week 0 at Week 4 | -0.09 (0.31) | -0.16 (0.50) | 0.04 (0.43)
  Change from Week 0 at Week 6: number analyzed (Participants) | 15 | 18 | 17
  Change from Week 0 at Week 6 | -0.05 (0.48) | -0.16 (0.69) | 0.05 (0.46)

4. Secondary Outcome: Scale for the Assessment of Negative Symptoms (SANS) - Anhedonia
Description: Mean score by treatment and week. Scores range from 0-5, with higher scores indicating a worse outcome.
Time Frame: Every other week for 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1: Oxytocin/Placebo-galantamine | 2: Galantamine/Placebo-oxytocin | 3: Placebo-galantamine /Placebo-oxytocin
Number analyzed (Participants) | 15 | 19 | 19
units on a scale
  Treatment Week 0 | 2.42 (0.59) | 2.60 (0.80) | 2.66 (0.69)
  Treatment Week 2 | 2.42 (0.64) | 2.59 (0.86) | 2.58 (0.66)
  Treatment Week 4: number analyzed (Participants) | 15 | 18 | 18
  Treatment Week 4 | 2.27 (0.78) | 2.46 (0.99) | 2.60 (0.64)
  Treatment Week 6: number analyzed (Participants) | 15 | 18 | 17
  Treatment Week 6 | 2.33 (0.49) | 2.43 (0.98) | 2.66 (0.60)
  Change from Week 0 at Week 2 | 0.00 (0.37) | -0.01 (0.40) | -0.08 (0.51)
  Change from Week 0 at Week 4: number analyzed (Participants) | 15 | 18 | 18
  Change from Week 0 at Week 4 | -0.15 (0.68) | -0.11 (.013) | 0.01 (0.50)
  Change from Week 0 at Week 6: number analyzed (Participants) | 15 | 18 | 17
  Change from Week 0 at Week 6 | -0.09 (0.38) | -0.14 (0.38) | 0.12 (0.47)

5. Secondary Outcome: Scale for the Assessment of Negative Symptoms (SANS) - Alogia
Description: Mean score by treatment and week. Scores range from 0-5, with higher scores indicating a worse outcome.
Time Frame: Every other week for 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1: Oxytocin/Placebo-galantamine | 2: Galantamine/Placebo-oxytocin | 3: Placebo-galantamine /Placebo-oxytocin
Number analyzed (Participants) | 15 | 19 | 19
units on a scale
  Treatment Week 0 | 0.60 (0.61) | 0.95 (0.65) | 0.99 (0.69)
  Treatment Week 2 | 0.44 (0.67) | 0.89 (0.59) | 0.89 (0.80)
  Treatment Week 4: number analyzed (Participants) | 15 | 18 | 18
  Treatment Week 4 | 0.56 (0.70) | 0.85 (0.50) | 0.80 (0.61)
  Treatment Week 6: number analyzed (Participants) | 15 | 18 | 17
  Treatment Week 6 | 0.56 (0.69) | 0.78 (0.44) | 0.69 (0.57)
  Change from Week 0 at Week 2 | -0.16 (0.42) | -0.05 (0.36) | -0.10 (0.35)
  Change from Week 0 at Week 4: number analyzed (Participants) | 15 | 18 | 18
  Change from Week 0 at Week 4 | -0.04 (0.41) | -0.03 (0.37) | -0.17 (0.31)
  Change from Week 0 at Week 6: number analyzed (Participants) | 15 | 18 | 17
  Change from Week 0 at Week 6 | -0.04 (0.46) | -0.10 (0.31) | -0.19 (0.31)

6. Secondary Outcome: Scale for the Assessment of Negative Symptoms (SANS) - Blunted Affect
Description: Mean score by treatment and week. Scores range from 0-5, with higher scores indicating a worse outcome.
Time Frame: Every other week for 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1: Oxytocin/Placebo-galantamine | 2: Galantamine/Placebo-oxytocin | 3: Placebo-galantamine /Placebo-oxytocin
Number analyzed (Participants) | 15 | 19 | 19
units on a scale
  Treatment Week 0 | 1.67 (0.86) | 1.96 (1.06) | 2.21 (0.97)
  Treatment Week 2 | 1.32 (0.90) | 1.89 (1.10) | 2.05 (1.12)
  Treatment Week 4: number analyzed (Participants) | 15 | 18 | 18
  Treatment Week 4 | 1.52 (0.91) | 1.79 (0.99) | 1.94 (0.98)
  Treatment Week 6: number analyzed (Participants) | 15 | 18 | 17
  Treatment Week 6 | 1.48 (0.96) | 1.70 (1.05) | 1.85 (0.94)
  Change from Week 0 at Week 2 | -0.35 (0.36) | -0.07 (0.36) | -0.16 (0.47)
  Change from Week 0 at Week 4: number analyzed (Participants) | 15 | 18 | 18
  Change from Week 0 at Week 4 | -0.15 (0.44) | -0.09 (0.33) | -0.19 (0.60)
  Change from Week 0 at Week 6: number analyzed (Participants) | 15 | 18 | 17
  Change from Week 0 at Week 6 | -0.19 (0.36) | -0.17 (0.40) | -0.19 (0.38)

7. Secondary Outcome: Brief Psychiatric Rating Scale (BPRS) - Total Score
Description: The total BPRS score is calculated by adding the scores for scales #1-#18. Each scale ranges from "1=Not Present" to "7=Very Severe". Total scores range from a minimum score of 18 to a maximum score of 126. A higher total score indicates a more severe psychiatric symptom rating.
Time Frame: Every other week for 6 weeks
Population: Safety data available for 56 participants exposed to study treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1: Oxytocin/Placebo-galantamine | 2: Galantamine/Placebo-oxytocin | 3: Placebo-galantamine /Placebo-oxytocin
Number analyzed (Participants) | 16 | 20 | 20
units on a scale
  Treatment Week 0 | 34.16 (5.66) | 30.35 (6.66) | 32.65 (7.09)
  Treatment Week 2: number analyzed (Participants) | 15 | 19 | 20
  Treatment Week 2 | 34.00 (7.46) | 28.95 (7.83) | 31.75 (7.26)
  Treatment Week 4: number analyzed (Participants) | 15 | 18 | 18
  Treatment Week 4 | 34.07 (6.15) | 27.83 (6.88) | 31.72 (7.25)
  Treatment Week 6: number analyzed (Participants) | 15 | 18 | 17
  Treatment Week 6 | 34.33 (5.09) | 27.67 (6.42) | 32.18 (6.21)

8. Secondary Outcome: Brief Psychiatric Rating Scale (BPRS) - Psychosis Score
Description: The psychosis score is calculated by adding the scores for scales #4 Conceptual Disorganization, #11 Suspiciousness, #12 Hallucinatory Behavior, and #15 Unusual Thought Content. Each scale ranges from "1=Not Present" to "7=Very Severe". The minimum psychosis score is 4 and the maximum psychosis score is 28. A higher score indicates a more severe psychosis rating.
Time Frame: Every other week for 6 weeks
Population: Safety data available for the 56 participants exposed to study treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 16 | 20 | 20
units on a scale
  Treatment Week 0 | 9.34 (3.20) | 7.30 (3.01) | 8.18 (3.80)
  Treatment Week 2: number analyzed (Participants) | 15 | 19 | 20
  Treatment Week 2 | 9.40 (3.79) | 7.21 (3.61) | 7.90 (3.86)
  Treatment Week 4: number analyzed (Participants) | 15 | 18 | 18
  Treatment Week 4 | 9.87 (3.60) | 7.00 (3.48) | 8.06 (4.09)
  Treatment Week 6: number analyzed (Participants) | 15 | 18 | 17
  Treatment Week 6 | 9.67 (2.87) | 6.78 (3.21) | 7.59 (4.35)

9. Secondary Outcome: Calgary Depression Scale (CDS) - Total Score
Description: Total score calculated by adding scores for scales #1-#9. Each scale ranges from "0=Absent" to "3=Severe". The minimum total CDS score is 0 and the maximum total CDS score is 27. A higher score indicates a more severe depression rating.
Time Frame: Every other week for 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1: Oxytocin/Placebo-galantamine | 2: Galantamine/Placebo-oxytocin | 3: Placebo-galantamine /Placebo-oxytocin
Number analyzed (Participants) | 15 | 19 | 19
units on a scale
  Treatment Week 0 | 2.37 (2.70) | 0.84 (1.07) | 1.59 (1.54)
  Treatment Week 2 | 2.20 (2.54) | 1.05 (1.65) | 1.00 (1.29)
  Treatment Week 4: number analyzed (Participants) | 15 | 18 | 18
  Treatment Week 4 | 2.13 (2.13) | 0.67 (1.28) | 0.94 (1.97)
  Treatment Week 6: number analyzed (Participants) | 15 | 18 | 17
  Treatment Week 6 | 1.67 (2.47) | 0.50 (0.71) | 1.29 (1.45)

10. Secondary Outcome: Arizona Sexual Experience Questionnaire (ASEX) Female
Description: Mean ASEX total scores by treatment and week for female participants. Total scores are calculated by adding scores for scales #1-#5. Each scale ranges from "1=Easily/Extremely" to "6=Never/None". The minimum total ASEX score is 5 and the maximum score is 30. Lower scores indicate more positive sexual experiences.
Time Frame: Once during evaluation and once at the end of 6 weeks of study treatment
Population: Female participants who completed at least two weeks follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1: Oxytocin/Placebo-galantamine | 2: Galantamine/Placebo-oxytocin | 3: Placebo-galantamine /Placebo-oxytocin
Number analyzed (Participants) | 2 | 6 | 3
units on a scale
  Treatment Week 0 | 10.5 (0.7) | 21.2 (7.6) | 29.0 (1.7)
  Treatment Week 6: number analyzed (Participants) | 2 | 6 | 2
  Treatment Week 6 | 13.5 (0.7) | 19.2 (9.3) | 30.0 (0)
  Change: number analyzed (Participants) | 2 | 6 | 2
  Change | 3.0 (0.0) | -2.0 (3.5) | 0.0 (0.0)

11. Secondary Outcome: Arizona Sexual Experience Questionnaire (ASEX) Male
Description: Mean ASEX total scores by treatment and week for male participants. Total scores are calculated by adding scores for scales #1-#5. Total scores are calculated by adding scores for scales #1-#5. Each scale ranges from "1=Easily/Extremely" to "6=Never/None". The minimum total ASEX score is 5 and the maximum score is 30. Lower scores indicate more positive sexual experiences.
Time Frame: Once during evaluation and once at the end of 6 weeks of study treatment
Population: Male participants who completed at least two weeks follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1: Oxytocin/Placebo-galantamine | 2: Galantamine/Placebo-oxytocin | 3: Placebo-galantamine /Placebo-oxytocin
Number analyzed (Participants) | 14 | 14 | 16
units on a scale
  Treatment Week 0: number analyzed (Participants) | 13 | 14 | 16
  Treatment Week 0 | 16.5 (9.2) | 18.1 (6.7) | 20.8 (6.3)
  Treatment Week 6: number analyzed (Participants) | 14 | 12 | 13
  Treatment Week 6 | 17.1 (8.5) | 20.2 (7.5) | 21.7 (7.7)
  Change: number analyzed (Participants) | 14 | 12 | 12
  Change | 1.5 (7.8) | 1.6 (5.0) | 0.8 (6.2)

12. Secondary Outcome: Vital Signs - Diastolic Blood Pressure
Description: Mean diastolic blood pressure by treatment and follow-up week
Time Frame: Weekly for 6 weeks
Population: Safety data for 56 participants exposed to study treatment.
Measure: Mean (Standard Deviation); unit: mm-Hg
Arm/Group | 1: Oxytocin/Placebo-galantamine | 2: Galantamine/Placebo-oxytocin | 3: Placebo-galantamine /Placebo-oxytocin
Number analyzed (Participants) | 16 | 20 | 20
mm-Hg
  Treatment Week 0 | 78.8 (8.3) | 76.6 (10.7) | 78.3 (10.1)
  Treatment Week 1: number analyzed (Participants) | 15 | 19 | 19
  Treatment Week 1 | 78.4 (9.0) | 76.2 (8.9) | 75.5 (10.8)
  Treatment Week 2: number analyzed (Participants) | 15 | 19 | 19
  Treatment Week 2 | 76.7 (9.1) | 77.5 (8.4) | 79.7 (10.6)
  Treatment Week 3: number analyzed (Participants) | 15 | 16 | 19
  Treatment Week 3 | 75.0 (10.6) | 79.1 (6.9) | 78.9 (8.1)
  Treatment Week 4: number analyzed (Participants) | 15 | 18 | 18
  Treatment Week 4 | 73.9 (8.2) | 75.1 (7.3) | 73.7 (9.7)
  Treatment Week 5: number analyzed (Participants) | 15 | 16 | 17
  Treatment Week 5 | 76.2 (8.8) | 79.2 (8.4) | 77.2 (10.9)
  Treatment Week 6: number analyzed (Participants) | 15 | 18 | 17
  Treatment Week 6 | 74.4 (8.3) | 80.7 (6.9) | 76.0 (9.9)

13. Secondary Outcome: Vital Signs - Systolic Blood Pressure
Description: Mean systolic blood pressure by treatment and follow-up week
Time Frame: Weekly for 6 weeks
Population: Safety data for 56 participants exposed to study treatment.
Measure: Mean (Standard Deviation); unit: mm-Hg
Arm/Group | 1: Oxytocin/Placebo-galantamine | 2: Galantamine/Placebo-oxytocin | 3: Placebo-galantamine /Placebo-oxytocin
Number analyzed (Participants) | 16 | 20 | 20
mm-Hg
  Treatment Week 0 | 128.4 (16.7) | 123.4 (17.3) | 132.3 (19.6)
  Treatment Week 1: number analyzed (Participants) | 15 | 19 | 19
  Treatment Week 1 | 126.1 (16.9) | 123.9 (15.0) | 127.4 (22.1)
  Treatment Week 2: number analyzed (Participants) | 15 | 19 | 19
  Treatment Week 2 | 121.9 (20.5) | 123.7 (13.8) | 136.2 (25.1)
  Treatment Week 3: number analyzed (Participants) | 15 | 16 | 19
  Treatment Week 3 | 129.5 (21.1) | 127.3 (19.0) | 137.7 (17.0)
  Treatment Week 4: number analyzed (Participants) | 15 | 18 | 18
  Treatment Week 4 | 124.8 (17.3) | 123.8 (19.0) | 129.9 (16.5)
  Treatment Week 5: number analyzed (Participants) | 15 | 16 | 17
  Treatment Week 5 | 128.4 (20.5) | 126.9 (20.1) | 132.8 (19.5)
  Treatment Week 6: number analyzed (Participants) | 15 | 18 | 17
  Treatment Week 6 | 124.0 (17.5) | 129.6 (16.1) | 134.5 (19.4)

14. Secondary Outcome: Vital Signs - Weight
Description: Mean weight (kg) by treatment and follow-up week
Time Frame: Weekly for 6 weeks
Population: Safety data for 56 participants exposed to study treatment.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | 1: Oxytocin/Placebo-galantamine | 2: Galantamine/Placebo-oxytocin | 3: Placebo-galantamine /Placebo-oxytocin
Number analyzed (Participants) | 16 | 20 | 20
kg
  Treatment Week 0 | 96.5 (18.4) | 96.2 (16.2) | 96.4 (20.0)
  Treatment Week 1: number analyzed (Participants) | 15 | 19 | 18
  Treatment Week 1 | 97.8 (19.1) | 97.5 (16.0) | 97.9 (18.9)
  Treatment Week 2: number analyzed (Participants) | 15 | 19 | 19
  Treatment Week 2 | 98.0 (18.9) | 97.5 (16.1) | 98.3 (18.8)
  Treatment Week 3: number analyzed (Participants) | 15 | 16 | 19
  Treatment Week 3 | 98.0 (18.9) | 94.5 (13.8) | 98.4 (19.5)
  Treatment Week 4: number analyzed (Participants) | 14 | 18 | 18
  Treatment Week 4 | 100.0 (17.9) | 95.5 (14.4) | 100.3 (17.7)
  Treatment Week 5: number analyzed (Participants) | 15 | 16 | 17
  Treatment Week 5 | 98.1 (18.6) | 94.0 (14.6) | 100.8 (17.7)
  Treatment Week 6: number analyzed (Participants) | 15 | 18 | 17
  Treatment Week 6 | 97.6 (18.0) | 95.1 (14.7) | 97.9 (16.3)

15. Secondary Outcome: Vital Signs - Pulse
Description: Mean sitting pulse (bpm) by treatment and follow-up week
Time Frame: Weekly for 6 weeks
Population: Safety data for 56 participants exposed to study treatment.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | 1: Oxytocin/Placebo-galantamine | 2: Galantamine/Placebo-oxytocin | 3: Placebo-galantamine /Placebo-oxytocin
Number analyzed (Participants) | 16 | 20 | 20
bpm
  Treatment Week 0 | 81.2 (10.4) | 86.0 (14.1) | 85.2 (13.4)
  Treatment Week 1: number analyzed (Participants) | 15 | 19 | 19
  Treatment Week 1 | 86.2 (18.8) | 91.6 (14.9) | 89.3 (16.7)
  Treatment Week 2: number analyzed (Participants) | 15 | 19 | 19
  Treatment Week 2 | 82.7 (17.3) | 91.3 (14.2) | 87.3 (15.3)
  Treatment Week 3: number analyzed (Participants) | 15 | 16 | 19
  Treatment Week 3 | 76.5 (11.5) | 89.2 (15.6) | 89.2 (13.8)
  Treatment Week 4: number analyzed (Participants) | 15 | 18 | 18
  Treatment Week 4 | 79.6 (13.2) | 88.6 (12.9) | 83.7 (14.2)
  Treatment Week 5: number analyzed (Participants) | 15 | 16 | 17
  Treatment Week 5 | 78.4 (13.2) | 98.6 (28.1) | 90.5 (16.0)
  Treatment Week 6: number analyzed (Participants) | 15 | 18 | 17
  Treatment Week 6 | 76.1 (15.0) | 85.2 (16.6) | 84.7 (12.2)

16. Secondary Outcome: Simpson-Angus Scale (SAS)
Description: SAS total score for extrapyramidal side effects: Frequencies of greatest within-participant increase (worsening) from pre-treatment baseline, by treatment group. Total scores calculated by adding scores from scales #1-#11. Each scale ranges from "0=None/Normal" to "4=Extreme/Severe". The minimum total score is 0 and the maximum score is 44. Higher scores indicate a more severe extrapyramidal side effect rating.
Time Frame: Baseline, week 3, and week 6
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | 1: Oxytocin/Placebo-galantamine | 2: Galantamine/Placebo-oxytocin | 3: Placebo-galantamine /Placebo-oxytocin
Number analyzed (Participants) | 15 | 19 | 19
percentage of participants
  No worsening (0) | 80 | 63.16 | 78.95
  Worsening of 1 | 16.67 | 10.53 | 10.53
  Worsening of 2 | 6.67 | 15.79 | 0
  Worsening of 3 | 6.67 | 5.26 | 5.26
  Worsening of 4 | 0 | 5.26 | 0
  Worsening of 10 | 0 | 0 | 5.26

17. Secondary Outcome: Abnormal Involuntary Movement Scale (AIMS)
Description: AIMS Total Score: Frequencies of Maximum Within- Participant Increases (worsening) from Baseline by Treatment Group. Total score calculated by adding scores from scales #1-#10. Each scale ranges from "0=None" to "4=Severe". The minimum total AIMS score is 0 and the maximum score is 40. Higher scores indicate a more severe abnormal involuntary movement rating.
Time Frame: Treatment Week 0 and Week 6
Population: 50 participants who completed the trial.
Measure: Number; unit: percentage of participants
Arm/Group | 1: Oxytocin/Placebo-galantamine | 2: Galantamine/Placebo-oxytocin | 3: Placebo-galantamine /Placebo-oxytocin
Number analyzed (Participants) | 15 | 18 | 17
percentage of participants
  No worsening (0) | 86.67 | 77.78 | 76.47
  Worsening of 1 | 6.67 | 16.67 | 17.65
  Worsening of 2 | 6.67 | 0 | 0
  Worsening of 3 | 0 | 0 | 5.88
  Worsening of 5 | 0 | 5.56 | 0

18. Secondary Outcome: Electrocardiogram (EKG)
Description: Mean corrected QT interval (QTc) by study week and treatment.
Time Frame: Once during Evaluation and once at Treatment Week 6
Population: 50 participants who completed the trial.
Measure: Mean (Standard Deviation); unit: QTc
Arm/Group | 1: Oxytocin/Placebo-galantamine | 2: Galantamine/Placebo-oxytocin | 3: Placebo-galantamine /Placebo-oxytocin
Number analyzed (Participants) | 15 | 18 | 17
QTc
  Evaluation Week 0: number analyzed (Participants) | 14 | 17 | 17
  Evaluation Week 0 | 416.5 (23.1) | 419.0 (26.6) | 422.6 (25.5)
  Treatment Week 6: number analyzed (Participants) | 15 | 18 | 16
  Treatment Week 6 | 415.7 (28.3) | 408.1 (27.2) | 423.8 (26.7)
  Change: number analyzed (Participants) | 14 | 17 | 16
  Change | -2.9 (20.7) | -10.2 (18.3) | 0.9 (20.3)

19. Secondary Outcome: Barnes Akathisia Scale (BAS) - Global Score
Description: For each subject, the largest increase from baseline in the global akathisia score at any visit during follow-up was calculated. The global akathisia score ranges from "0=Absent" to "5=Severe Akathisia". Higher scores indicate a more severe global rating of akathisia.
Time Frame: Treatment Week 0 and Week 6
Population: 50 participants who completed the trial.
Measure: Number; unit: percentage of participants
Arm/Group | 1: Oxytocin/Placebo-galantamine | 2: Galantamine/Placebo-oxytocin | 3: Placebo-galantamine /Placebo-oxytocin
Number analyzed (Participants) | 15 | 18 | 17
percentage of participants
  No worsening (0) | 93.33 | 100 | 94.12
  Worsening of 1 | 6.67 | 0 | 5.88

20. Secondary Outcome: Blood Oxytocin Levels
Description: Blood Oxytocin Levels by Treatment and Visit
Time Frame: Treatment Week 0 and Week 6
Population: Of the 56 participants exposed to study drug, 3 withdrew before any efficacy data was collected, leaving 53 for whom at least some interim efficacy data was collected.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | 1: Oxytocin/Placebo-galantamine | 2: Galantamine/Placebo-oxytocin | 3: Placebo-galantamine /Placebo-oxytocin
Number analyzed (Participants) | 16 | 20 | 17
pg/mL
  Treatment Week 0 | 18.22 (15.52) | 13.76 (6.96) | 14.69 (7.99)
  Treatment Week 6: number analyzed (Participants) | 14 | 15 | 13
  Treatment Week 6 | 17.22 (17.02) | 10.11 (3.42) | 13.21 (9.32)
  Change: number analyzed (Participants) | 14 | 15 | 11
  Change | -1.88 (14.09) | -2.99 (5.2) | -1.73 (3.95)

21. Secondary Outcome: Laboratory Measures - ALT/SGPT
Description: Alanine transaminase/serum glutamic-pyruvic transaminase (ALT/SGPT) blood levels by treatment group and visit.
Time Frame: Once during evaluation and once at the end of 6 weeks of study treatment
Population: Available participant lab data at Evaluation and Week 6.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | 1: Oxytocin/Placebo-galantamine | 2: Galantamine/Placebo-oxytocin | 3: Placebo-galantamine /Placebo-oxytocin
Number analyzed (Participants) | 15 | 20 | 20
U/L
  Evaluation: number analyzed (Participants) | 15 | 19 | 20
  Evaluation | 22.87 (8.68) | 31.26 (22.93) | 27.40 (19.78)
  Treatment Week 6: number analyzed (Participants) | 15 | 20 | 19
  Treatment Week 6 | 20.67 (13.03) | 28.90 (22.81) | 27.74 (16.62)
  Change: number analyzed (Participants) | 13 | 17 | 16
  Change | -2.15 (10.20) | -2.65 (6.14) | 0.31 (8.10)

22. Secondary Outcome: Laboratory Measures - AST/SGOT
Description: Aspartate aminotransferase/serum glutamic oxaloacetic transaminase (AST/SGOT) blood levels by treatment group and visit.
Time Frame: Once during evaluation and once at the end of 6 weeks of study treatment
Population: Available participant lab data at Evaluation and Week 6.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | 1: Oxytocin/Placebo-galantamine | 2: Galantamine/Placebo-oxytocin | 3: Placebo-galantamine /Placebo-oxytocin
Number analyzed (Participants) | 15 | 20 | 20
U/L
  Evaluation: number analyzed (Participants) | 15 | 19 | 20
  Evaluation | 19.87 (5.46) | 22.68 (9.68) | 22.50 (9.29)
  Treatment Week 6: number analyzed (Participants) | 15 | 20 | 19
  Treatment Week 6 | 20.27 (8.94) | 21.45 (10.16) | 23.58 (9.26)
  Change: number analyzed (Participants) | 13 | 17 | 16
  Change | -1.46 (4.20) | -1.53 (8.13) | 1.00 (5.43)

23. Secondary Outcome: Laboratory Measures - Alkaline Phosphatase
Description: Alkaline phosphatase blood level by treatment group and visit.
Time Frame: Once during evaluation and once at the end of 6 weeks of study treatment
Population: Available participant lab data at Evaluation at Week 6.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | 1: Oxytocin/Placebo-galantamine | 2: Galantamine/Placebo-oxytocin | 3: Placebo-galantamine /Placebo-oxytocin
Number analyzed (Participants) | 15 | 20 | 20
U/L
  Evaluation: number analyzed (Participants) | 15 | 19 | 20
  Evaluation | 83.47 (21.56) | 83.42 (16.29) | 86.40 (23.37)
  Treatment Week 6: number analyzed (Participants) | 15 | 20 | 19
  Treatment Week 6 | 78.73 (31.09) | 82.50 (20.50) | 88.95 (29.67)
  Change: number analyzed (Participants) | 13 | 17 | 16
  Change | -4.77 (15.81) | 0.88 (10.29) | 1.19 (10.97)

24. Secondary Outcome: Laboratory Measures - Calcium
Description: Calcium blood levels by treatment group and visit.
Time Frame: Once during evaluation and once at the end of 6 weeks of study treatment
Population: Available participant lab data at Evaluation and Week 6.
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- 1: Oxytocin: Subjects randomized to oxytocin will receive oxytocin and placebo-galantamine
- 2: Galantamine: Subjects randomized to galantamine will receive galantamine and placebo-oxytocin
- 3: Placebo: Subjects randomized to placebo will receive placebo-galantamine and placebo-oxytocin
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 15 | 20 | 20
mg/dL
  Evaluation: number analyzed (Participants) | 15 | 19 | 20
  Evaluation | 9.53 (0.33) | 9.36 (0.31) | 9.58 (0.41)
  Treatment Week 6: number analyzed (Participants) | 15 | 20 | 19
  Treatment Week 6 | 9.57 (0.32) | 9.23 (0.31) | 9.54 (0.44)
  Change: number analyzed (Participants) | 13 | 17 | 16
  Change | 0.12 (0.33) | -0.16 (0.21) | -0.03 (0.36)

25. Secondary Outcome: Laboratory Measures - Sodium
Description: Sodium blood levels by treatment group and visit.
Time Frame: Once during evaluation and once at the end of 6 weeks of study treatment
Population: Available participant lab data at Evaluation and Week 6.
Measure: Mean (Standard Deviation); unit: mE/qL
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 15 | 20 | 20
mE/qL
  Evaluation: number analyzed (Participants) | 15 | 19 | 20
  Evaluation | 138.53 (2.29) | 139.53 (2.89) | 137.30 (4.28)
  Treatment Week 6: number analyzed (Participants) | 15 | 20 | 19
  Treatment Week 6 | 138.53 (3.02) | 139.15 (2.16) | 137.47 (3.96)
  Change: number analyzed (Participants) | 13 | 17 | 16
  Change | 0.15 (1.63) | -0.53 (3.22) | 0.31 (2.82)

26. Secondary Outcome: Laboratory Measures - Potassium
Description: Potassium blood levels by treatment group and visit.
Time Frame: Once during evaluation and once at the end of 6 weeks of study treatment
Population: Available participant lab data at Evaluation and Week 6.
Measure: Mean (Standard Deviation); unit: mE/qL
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 15 | 20 | 20
mE/qL
  Evaluation: number analyzed (Participants) | 15 | 19 | 20
  Evaluation | 4.20 (0.47) | 4.14 (0.31) | 4.17 (0.28)
  Treatment Week 6: number analyzed (Participants) | 15 | 20 | 19
  Treatment Week 6 | 4.07 (0.32) | 4.01 (0.27) | 4.16 (0.39)
  Change: number analyzed (Participants) | 13 | 17 | 16
  Change | -0.12 (0.43) | -0.15 (0.22) | 0.00 (0.31)

27. Secondary Outcome: Laboratory Measures - Chloride
Description: Chloride blood levels by treatment group and visit.
Time Frame: Once during evaluation and once at the end of 6 weeks of study treatment
Population: Available participant lab data for Evaluation and Week 6.
Measure: Mean (Standard Deviation); unit: mE/qL
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 15 | 20 | 20
mE/qL
  Evaluation: number analyzed (Participants) | 15 | 19 | 20
  Evaluation | 100.60 (2.95) | 102.79 (3.41) | 100.15 (4.21)
  Treatment Week 6: number analyzed (Participants) | 15 | 20 | 19
  Treatment Week 6 | 101.53 (3.54) | 102.90 (2.63) | 100.47 (3.78)
  Change: number analyzed (Participants) | 13 | 17 | 16
  Change | 0.62 (1.89) | -0.06 (2.70) | 0.56 (2.80)

28. Secondary Outcome: Laboratory Measures - CO2
Description: Carbon Dioxide (CO2) blood levels by treatment group and visit.
Time Frame: Once during evaluation and once at the end of 6 weeks of study treatment
Population: Available participant lab data for Evaluation and Week 6.
Measure: Mean (Standard Deviation); unit: mE/qL
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 15 | 20 | 20
mE/qL
  Evaluation: number analyzed (Participants) | 15 | 19 | 20
  Evaluation | 23.47 (2.13) | 22.42 (3.01) | 23.40 (2.52)
  Treatment Week 6: number analyzed (Participants) | 15 | 20 | 18
  Treatment Week 6 | 23.27 (2.09) | 22.50 (2.33) | 22.83 (2.15)
  Change: number analyzed (Participants) | 13 | 17 | 15
  Change | -0.31 (2.21) | -0.06 (2.77) | -0.20 (1.52)

29. Secondary Outcome: Laboratory Measures - Cholesterol
Description: Total cholesterol blood levels by treatment group and visit.
Time Frame: Once during evaluation and once at the end of 6 weeks of study treatment
Population: Available participant lab data for Evaluation and Week 6.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 14 | 15 | 15
mg/dL
  Evaluation: number analyzed (Participants) | 11 | 15 | 15
  Evaluation | 159.18 (19.18) | 166.07 (35.98) | 179.60 (37.43)
  Treatment Week 6: number analyzed (Participants) | 14 | 14 | 12
  Treatment Week 6 | 156.93 (22.57) | 162.93 (22.57) | 177.33 (36.76)
  Change: number analyzed (Participants) | 10 | 10 | 9
  Change | 1.50 (12.61) | -2.40 (15.87) | -11.44 (31.52)

30. Secondary Outcome: Laboratory Measures - HDL
Description: High-density lipoprotein (HDL) blood levels by treatment group and visit.
Time Frame: Once during evaluation and once at the end of 6 weeks of study treatment
Population: Available participant data from Evaluation and Week 6.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 13 | 14 | 14
mg/dL
  Evaluation: number analyzed (Participants) | 11 | 14 | 14
  Evaluation | 44.09 (12.31) | 45.50 (14.43) | 41.14 (10.17)
  Treatment Week 6: number analyzed (Participants) | 13 | 14 | 12
  Treatment Week 6 | 44.31 (14.07) | 43.64 (11.62) | 41.42 (10.75)
  Change: number analyzed (Participants) | 10 | 9 | 9
  Change | -0.70 (6.31) | 2.11 (3.69) | -1.67 (4.50)

31. Secondary Outcome: Laboratory Measures - LDL
Description: Low-density lipoprotein (LDL) blood levels by treatment group and visit.
Time Frame: Once during evaluation and once at the end of 6 weeks of study treatment
Population: Available participant lab data for Evaluation and Week 6.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 13 | 14 | 14
mg/dL
  Evaluation: number analyzed (Participants) | 11 | 12 | 14
  Evaluation | 90.36 (25.02) | 91.25 (20.42) | 105.79 (37.30)
  Treatment Week 6: number analyzed (Participants) | 13 | 14 | 11
  Treatment Week 6 | 85.92 (28.72) | 92.29 (19.51) | 103.73 (33.32)
  Change: number analyzed (Participants) | 10 | 8 | 8
  Change | -0.60 (11.58) | -1.38 (14.92) | -13.00 (26.79)

32. Secondary Outcome: Laboratory Measures - Triglycerides
Description: Triglyceride blood levels by treatment group and visit.
Time Frame: Once during evaluation and once at the end of 6 weeks of study treatment
Population: Available participant lab data for Evaluation and Week 6.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 14 | 15 | 15
mg/dL
  Evaluation: number analyzed (Participants) | 11 | 15 | 15
  Evaluation | 124.55 (60.32) | 155.20 (118.82) | 163.47 (102.54)
  Treatment Week 6: number analyzed (Participants) | 14 | 14 | 12
  Treatment Week 6 | 124.79 (69.57) | 142.29 (99.53) | 162.17 (102.74)
  Change: number analyzed (Participants) | 10 | 10 | 9
  Change | 14.00 (40.14) | -39.30 (77.44) | 1.22 (49.85)

33. Secondary Outcome: Laboratory Measures - VLDL
Description: Very low density lipoprotein (VLDL) blood levels by treatment group and visit.
Time Frame: Once during evaluation and once at the end of 6 weeks of study treatment
Population: Available participant lab data for Evaluation and Week 6.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 12 | 13 | 12
mg/dL
  Evaluation: number analyzed (Participants) | 11 | 11 | 12
  Evaluation | 24.73 (12.04) | 22.00 (10.49) | 33.17 (22.59)
  Treatment Week 6: number analyzed (Participants) | 12 | 13 | 11
  Treatment Week 6 | 26.75 (13.93) | 23.62 (9.50) | 28.00 (14.04)
  Change: number analyzed (Participants) | 10 | 8 | 7
  Change | 2.80 (8.13) | -3.13 (6.31) | -0.43 (11.19)

34. Secondary Outcome: Laboratory Measures - Glucose
Description: Glucose blood levels by treatment group and visit.
Time Frame: Once during evaluation and once at the end of 6 weeks of study treatment
Population: Available participant lab data for Evaluation and Week 6.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 15 | 18 | 18
mg/dL
  Evaluation | 108.07 (47.12) | 98.61 (15.50) | 103.00 (21.86)
  Treatment Week 6: number analyzed (Participants) | 15 | 16 | 16
  Treatment Week 6 | 99.67 (19.53) | 102.13 (18.13) | 112.31 (33.36)
  Change: number analyzed (Participants) | 13 | 13 | 13
  Change | -9.23 (30.91) | 2.00 (20.64) | 9.77 (16.51)

35. Secondary Outcome: Laboratory Measures - Albumin
Description: Albumin blood levels by treatment group and visit.
Time Frame: Once during evaluation and once at the end of 6 weeks of study treatment
Population: Available participant lab data for Evaluation and Week 6.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 15 | 20 | 20
g/dL
  Evaluation: number analyzed (Participants) | 15 | 19 | 20
  Evaluation | 4.39 (0.24) | 4.27 (0.31) | 4.35 (0.30)
  Treatment Week 6: number analyzed (Participants) | 15 | 20 | 19
  Treatment Week 6 | 4.38 (0.25) | 4.23 (0.27) | 4.37 (0.32)
  Change: number analyzed (Participants) | 13 | 17 | 16
  Change | 0.04 (0.23) | -0.03 (0.35) | 0.03 (0.20)

36. Secondary Outcome: Laboratory Measures - Globulin
Description: Globulin blood levels by treatment group and visit.
Time Frame: Once during evaluation and once at the end of 6 weeks of study treatment
Population: Available participant lab data for Evaluation and Week 6.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 14 | 18 | 19
g/dL
  Evaluation: number analyzed (Participants) | 14 | 18 | 18
  Evaluation | 2.72 (0.40) | 2.81 (0.42) | 2.82 (0.37)
  Treatment Week 6 | 2.58 (0.54) | 2.66 (0.51) | 2.78 (0.38)
  Change: number analyzed (Participants) | 12 | 15 | 15
  Change | -0.15 (0.63) | -0.18 (0.38) | -0.09 (0.21)

37. Secondary Outcome: Laboratory Measures - A/G Ratio
Description: Albumin to Globulin (A/G) ratio in the blood by treatment group and visit.
Time Frame: Once during evaluation and once at the end of 6 weeks of study treatment
Population: Available participant date for Evaluation and Week 6.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 15 | 18 | 19
g/dL
  Evaluation: number analyzed (Participants) | 15 | 18 | 18
  Evaluation | 1.65 (0.29) | 1.58 (0.27) | 1.57 (0.26)
  Treatment Week 6: number analyzed (Participants) | 13 | 17 | 19
  Treatment Week 6 | 1.71 (0.64) | 1.62 (0.31) | 1.60 (0.26)
  Change: number analyzed (Participants) | 12 | 14 | 15
  Change | 0.04 (0.22) | 0.05 (0.18) | 0.07 (0.12)

38. Secondary Outcome: Laboratory Measures - Bilirubin
Description: Bilirubin blood level by treatment group and visit.
Time Frame: Once during evaluation and once at the end of 6 weeks of study treatment
Population: Available participant data for Evaluation and Week 6.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 15 | 20 | 19
mg/dL
  Evaluation: number analyzed (Participants) | 15 | 19 | 19
  Evaluation | 0.45 (0.29) | 0.35 (0.19) | 0.40 (0.26)
  Treatment Week 6 | 0.49 (0.24) | 0.39 (0.24) | 0.38 (0.15)
  Change: number analyzed (Participants) | 13 | 17 | 15
  Change | 0.03 (0.13) | 0.05 (0.23) | 0.03 (0.13)

39. Secondary Outcome: Laboratory Measures - Protein
Description: Protein blood level by treatment group and visit.
Time Frame: Once during evaluation and once at the end of 6 weeks of study treatment
Population: Available participant data for Evaluation and Week 6.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 15 | 20 | 20
g/dL
  Evaluation: number analyzed (Participants) | 15 | 19 | 20
  Evaluation | 7.10 (0.32) | 7.07 (0.41) | 7.17 (0.40)
  Treatment Week 6: number analyzed (Participants) | 15 | 20 | 19
  Treatment Week 6 | 7.14 (0.42) | 6.92 (0.45) | 7.15 (0.42)
  Change: number analyzed (Participants) | 13 | 17 | 16
  Change | 0.07 (0.30) | -0.13 (0.34) | -0.04 (0.37)

40. Secondary Outcome: Laboratory Measures - BUN
Description: BUN blood level by treatment group and visit.
Time Frame: Once during evaluation and once at the end of 6 weeks of study treatment
Population: Available participant data for Evaluation and Week 6.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 15 | 20 | 20
mg/dL
  Evaluation: number analyzed (Participants) | 15 | 19 | 20
  Evaluation | 12.80 (4.92) | 10.74 (3.18) | 11.95 (4.10)
  Treatment Week 6: number analyzed (Participants) | 15 | 20 | 19
  Treatment Week 6 | 12.73 (4.85) | 11.55 (3.41) | 12.00 (4.76)
  Change: number analyzed (Participants) | 13 | 17 | 16
  Change | 0.15 (2.82) | 1.06 (3.07) | -0.06 (3.38)

41. Secondary Outcome: Side Effect Checklist (SEC) - Abdominal Pain
Description: Percentage of participants with new onset or worsening compared to baseline of "Abdominal Pain" rating on the SEC, by Treatment Group.
Time Frame: Weekly for 6 weeks
Population: Safety data for 56 participants exposed to study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 16 | 20 | 20
percentage of participants | 12.5 | 5.0 | 10.0

42. Secondary Outcome: Side Effect Checklist (SEC) - Anorexia
Description: Percentage of participants with new onset or worsening compared to baseline of "Anorexia" rating on the SEC, by Treatment Group.
Time Frame: Weekly for 6 weeks
Population: Safety data for 56 participants exposed to study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 16 | 20 | 20
percentage of participants | 18.8 | 10.0 | 15.0

43. Secondary Outcome: Side Effect Checklist (SEC) - Bruising Easily
Description: Percentage of participants with new onset or worsening compared to baseline of "Bruising Easily" rating on the SEC, by Treatment Group.
Time Frame: Weekly for 6 weeks
Population: Safety data for 56 participants exposed to study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 16 | 20 | 20
percentage of participants | 0.0 | 10.0 | 0.0

44. Secondary Outcome: Side Effect Checklist (SEC) - Constipation
Description: Percentage of participants with new onset or worsening compared to baseline of "Constipation" rating on the SEC, by Treatment Group.
Time Frame: Weekly for 6 weeks
Population: Safety data for 56 participants exposed to study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 16 | 20 | 20
percentage of participants | 0.0 | 0.0 | 0.0

45. Secondary Outcome: Side Effect Checklist (SEC) - Diarrhea
Description: Percentage of participants with new onset or worsening compared to baseline of "Diarrhea" rating on the SEC, by Treatment Group.
Time Frame: Weekly for 6 weeks
Population: Safety data for 56 participants exposed to study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 16 | 20 | 20
percentage of participants | 18.8 | 30.0 | 5.0

46. Secondary Outcome: Side Effect Checklist (SEC) - Dizziness
Description: Percentage of participants with new onset or worsening compared to baseline of "Dizziness" rating on the SEC, by Treatment Group.
Time Frame: Weekly for 6 weeks
Population: Safety data for 56 participants exposed to study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 16 | 20 | 20
percentage of participants | 18.8 | 30.0 | 5.0

47. Secondary Outcome: Side Effect Checklist (SEC) - Dry Eye
Description: Percentage of participants with new onset or worsening compared to baseline of "Dry Eye" rating on the SEC, by Treatment Group.
Time Frame: Weekly for 6 weeks
Population: Safety data for 56 participants exposed to study treatment minus 6 participants who had missing "dry eye" data.
Measure: Number; unit: percentage of participants
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 15 | 18 | 17
percentage of participants | 6.7 | 0.0 | 5.9

48. Secondary Outcome: Side Effect Checklist (SEC) - Dry Mouth
Description: Percentage of participants with new onset or worsening compared to baseline of "Dry Mouth" rating on the SEC, by Treatment Group.
Time Frame: Weekly for 6 weeks
Population: Safety data for 56 participants exposed to study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 16 | 20 | 20
percentage of participants | 18.8 | 5.0 | 10.0

49. Secondary Outcome: Side Effect Checklist (SEC) - Enuresis
Description: Percentage of participants with new onset or worsening compared to baseline of "Enuresis" rating on the SEC, by Treatment Group.
Time Frame: Weekly for 6 weeks
Population: Safety data for 56 participants exposed to study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 16 | 20 | 20
percentage of participants | 25.0 | 5.0 | 0.0

50. Secondary Outcome: Side Effect Checklist (SEC) - Excessive Tearing of the Eye
Description: Percentage of participants with new onset or worsening compared to baseline of "Excessive Tearing of the Eye" rating on the SEC, by Treatment Group.
Time Frame: Weekly for 6 weeks
Population: Safety data for 56 participants exposed to study treatment minus 6 participants who had missing "excessive tearing of the eye" data.
Measure: Number; unit: percentage of participants
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 15 | 18 | 17
percentage of participants | 6.7 | 5.6 | 5.9

51. Secondary Outcome: Side Effect Checklist (SEC) - Fever
Description: Percentage of participants with new onset or worsening compared to baseline of "Fever" rating on the SEC, by Treatment Group.
Time Frame: Weekly for 6 weeks
Population: Safety data for 56 participants exposed to study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 16 | 20 | 20
percentage of participants | 0.0 | 5.0 | 0.0

52. Secondary Outcome: Side Effect Checklist (SEC) - Headache
Description: Percentage of participants with new onset or worsening compared to baseline of "Headache" rating on the SEC, by Treatment Group.
Time Frame: Weekly for 6 weeks
Population: Safety data for 56 participants exposed to study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 16 | 20 | 20
percentage of participants | 12.5 | 25.0 | 15.0

53. Secondary Outcome: Side Effect Checklist (SEC) - Hyperhydrosis
Description: Percentage of participants with new onset or worsening compared to baseline of "Hyperhydrosis" rating on the SEC, by Treatment Group.
Time Frame: Weekly for 6 weeks
Population: Safety data for 56 participants exposed to study treatment minus 6 participants who had missing "Hyperhydrosis" data.
Measure: Number; unit: percentage of participants
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 15 | 18 | 17
percentage of participants | 0.0 | 0.0 | 0.0

54. Secondary Outcome: Side Effect Checklist (SEC) - Hypersalivation
Description: Percentage of participants with new onset or worsening compared to baseline of "Hypersalivation" rating on the SEC, by Treatment Group.
Time Frame: Weekly for 6 weeks
Population: Safety data for 56 participants exposed to study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 16 | 20 | 20
percentage of participants | 18.8 | 15.0 | 25.0

55. Secondary Outcome: Side Effect Checklist (SEC) - Insomnia
Description: Percentage of participants with new onset or worsening compared to baseline of "Insomnia" rating on the SEC, by Treatment Group.
Time Frame: Weekly for 6 weeks
Population: Safety data for 56 participants exposed to study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 16 | 20 | 20
percentage of participants | 18.8 | 10.0 | 5.0

56. Secondary Outcome: Side Effect Checklist (SEC) - Malaise
Description: Percentage of participants with new onset or worsening compared to baseline of "Malaise" rating on the SEC, by Treatment Group.
Time Frame: Weekly for 6 weeks
Population: Safety data for 56 participants exposed to study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 16 | 20 | 20
percentage of participants | 18.8 | 0.0 | 10.0

57. Secondary Outcome: Side Effect Checklist (SEC) - Mucosal Ulceration
Description: Percentage of participants with new onset or worsening compared to baseline of "Mucosal Ulceration" rating on the SEC, by Treatment Group.
Time Frame: Weekly for 6 weeks
Population: Safety data for 56 participants exposed to study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 16 | 20 | 20
percentage of participants | 6.3 | 5.0 | 0.0

58. Secondary Outcome: Side Effect Checklist (SEC) - Nasal Irritation
Description: Percentage of participants with new onset or worsening compared to baseline of "Nasal Irritation" rating on the SEC, by Treatment Group.
Time Frame: Weekly for 6 weeks
Population: Safety data for 56 participants exposed to study treatment minus 6 participants who had missing "nasal irritation" data.
Measure: Number; unit: percentage of participants
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 15 | 18 | 17
percentage of participants | 33.3 | 16.7 | 23.5

59. Secondary Outcome: Side Effect Checklist (SEC) - Nausea
Description: Percentage of participants with new onset or worsening compared to baseline of "Nausea" rating on the SEC, by Treatment Group.
Time Frame: Weekly for 6 weeks
Population: Safety data for 56 participants exposed to study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 16 | 20 | 20
percentage of participants | 18.8 | 15.0 | 5.0

60. Secondary Outcome: Side Effect Checklist (SEC) - Rash
Description: Percentage of participants with new onset or worsening compared to baseline of "Rash" rating on the SEC, by Treatment Group.
Time Frame: Weekly for 6 weeks
Population: Safety data for 56 participants exposed to study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 16 | 20 | 20
percentage of participants | 12.5 | 10.0 | 10.0

61. Secondary Outcome: Side Effect Checklist (SEC) - Restlessness
Description: Percentage of participants with new onset or worsening compared to baseline of "Restlessness" rating on the SEC, by Treatment Group.
Time Frame: Weekly for 6 weeks
Population: Safety data for 56 participants exposed to study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 16 | 20 | 20
percentage of participants | 18.8 | 10.0 | 15.0

62. Secondary Outcome: Side Effect Checklist (SEC) - Sedation
Description: Percentage of participants with new onset or worsening compared to baseline of "Sedation" rating on the SEC, by Treatment Group.
Time Frame: Weekly for 6 weeks
Population: Safety data for 56 participants exposed to study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 16 | 20 | 20
percentage of participants | 12.5 | 15.0 | 10.0

63. Secondary Outcome: Side Effect Checklist (SEC) - Sore Throat
Description: Percentage of participants with new onset or worsening compared to baseline of "Sore Throat" rating on the SEC, by Treatment Group.
Time Frame: Weekly for 6 weeks
Population: Safety data for 56 participants exposed to study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 16 | 20 | 20
percentage of participants | 6.3 | 10.0 | 5.0

64. Secondary Outcome: Side Effect Checklist (SEC) - Stiffness
Description: Percentage of participants with new onset or worsening compared to baseline of "Stiffness" rating on the SEC, by Treatment Group.
Time Frame: Weekly for 6 weeks
Population: Safety data for 56 participants exposed to study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 16 | 20 | 20
percentage of participants | 6.3 | 10.0 | 10.0

65. Secondary Outcome: Side Effect Checklist (SEC) - Tinnitus
Description: Percentage of participants with new onset or worsening compared to baseline of "Tinnitus" rating on the SEC, by Treatment Group.
Time Frame: Weekly for 6 weeks
Population: Safety data for 56 participants exposed to study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 16 | 20 | 19
percentage of participants | 0.0 | 0.0 | 10.5

66. Secondary Outcome: Side Effect Checklist (SEC) - Tremor
Description: Percentage of participants with new onset or worsening compared to baseline of "Tremor" rating on the SEC, by Treatment Group.
Time Frame: Weekly for 6 weeks
Population: Safety data for 56 participants exposed to study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 16 | 20 | 20
percentage of participants | 6.3 | 15.0 | 10.0

67. Secondary Outcome: Side Effect Checklist (SEC) - Urticaria
Description: Percentage of participants with new onset or worsening compared to baseline of "Urticaria" rating on the SEC, by Treatment Group.
Time Frame: Weekly for 6 weeks
Population: Safety data for 56 participants exposed to study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 16 | 20 | 20
percentage of participants | 18.8 | 15.0 | 15.0

68. Secondary Outcome: Side Effect Checklist (SEC) - Uterine Contractions
Description: Percentage of participants with new onset or worsening compared to baseline of "Uterine Contractions" rating on the SEC, by Treatment Group.
Time Frame: Weekly for 6 weeks
Population: Female participants
Measure: Number; unit: percentage of participants
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 2 | 6 | 3
percentage of participants | 0.0 | 0.0 | 0.0

69. Secondary Outcome: Side Effect Checklist (SEC) - Vomiting
Description: Percentage of participants with new onset or worsening compared to baseline of "Vomiting" rating on the SEC, by Treatment Group.
Time Frame: Weekly for 6 weeks
Population: Safety data for 56 participants exposed to study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 16 | 20 | 20
percentage of participants | 12.5 | 5.0 | 10.0

70. Secondary Outcome: Side Effect Checklist (SEC) - Weight Loss
Description: Percentage of participants with new onset or worsening compared to baseline of "Weight Loss" rating on the SEC, by Treatment Group.
Time Frame: Weekly for 6 weeks
Population: Safety data for 56 participants exposed to study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 16 | 20 | 20
percentage of participants | 18.8 | 5.0 | 25.0

71. Secondary Outcome: Side Effect Checklist (SEC) - Wheezing
Description: Percentage of participants with new onset or worsening compared to baseline of "Wheezing" rating on the SEC, by Treatment Group.
Time Frame: Weekly for 6 weeks
Population: Safety data for 56 participants exposed to study treatment minus 6 participants with missing "wheezing" data.
Measure: Number; unit: percentage of participants
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 15 | 18 | 17
percentage of participants | 13.3 | 5.6 | 11.8

72. Secondary Outcome: Neurocognitive Assessment Battery (MCCB) - Composite Score
Description: MCCB Composite Score by Week ranging from -10-100 with a higher score indicating a better outcome.
Time Frame: Once at Treatment Week 0 (baseline) and again at Treatment Week 6 (end of treatment).
Population: Cognitive data was collected at baseline and week 6, so only those participants who got to week 6 appear in cognitive outcome analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1: Oxytocin/Placebo-galantamine | 2: Galantamine/Placebo-oxytocin | 3: Placebo-galantamine /Placebo-oxytocin
Number analyzed (Participants) | 15 | 16 | 15
units on a scale
  Treatment Week 0 | 25.9 (13.0) | 24.5 (9.7) | 28.2 (9.6)
  Treatment Week 6 | 28.2 (14.1) | 26.2 (11.1) | 28.9 (11.8)
  Change | 2.3 (3.9) | 1.7 (4.0) | 0.7 (8.0)

73. Secondary Outcome: Neurocognitive Assessment Battery (MCCB) - Attention Vigilance
Description: MCCB Attention Vigilance domain score by week calculated from the Continuous Performance Test, Identical Pairs version. The domain score scale is 20-80, with higher scores indicating a better outcome.
  .
Time Frame: Once at Treatment Week 0 (baseline) and again at Treatment Week 6 (end of treatment).
Population: as for outcome 72
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 15 | 17 | 17
units on a scale
  Treatment Week 0 | 36.9 (8.8) | 33.5 (14.5) | 37.2 (10.9)
  Treatment Week 6 | 39.5 (11.3) | 34.5 (13.6) | 35.1 (12.7)
  Change | 2.6 (5.8) | 1.1 (6.9) | -2.1 (6.9)

74. Secondary Outcome: Neurocognitive Assessment Battery (MCCB) - Processing Speed
Description: MCCB Processing Speed domain score by week calculated from the Trail Making Test- Part A, Brief Assessment of Cognition in Schizophrenia- symbol coding subtest, and the Category fluency test- animal naming. The domain score scale is 20-80, with higher scores indicating a better outcome.
Time Frame: Once at Treatment Week 0 (baseline) and again at Treatment Week 6 (end of treatment).
Population: as for outcome 72
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 15 | 18 | 17
units on a scale
  Treatment Week 0 | 33.5 (13.1) | 31.9 (11.7) | 34.0 (10.9)
  Treatment Week 6 | 34.2 (11.6) | 35.4 (8.6) | 35.6 (12.7)
  Change | 0.7 (4.3) | 3.5 (5.6) | 1.6 (7.3)

75. Secondary Outcome: Neurocognitive Assessment Battery (MCCB) - Reasoning/Problem Solving
Description: MCCB Reasoning/Problem Solving domain score by week calculated from the Neuropsychological Assessment Battery- mazes subtest. The domain score scale is 20-80, with higher scores indicating a better outcome.
Time Frame: Once at Treatment Week 0 (baseline) and again at Treatment Week 6 (end of treatment).
Population: as for outcome 72
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 15 | 18 | 17
units on a scale
  Treatment Week 0 | 39.7 (10.8) | 39.3 (6.8) | 41.4 (8.4)
  Treatment Week 6 | 40.7 (9.4) | 42.9 (8.3) | 41.7 (9.7)
  Change | 1.0 (8.1) | 3.7 (5.1) | 0.3 (10.1)

76. Secondary Outcome: Neurocognitive Assessment Battery (MCCB) - Social Cognition
Description: MCCB Social Cognition domain score by week calculated from the Mayer-Salovey-Caruso Emotional Intelligence Test- managing emotions branch. The domain score scale is 20-80, with higher scores indicating a better outcome.
Time Frame: Once at Treatment Week 0 (baseline) and again at Treatment Week 6 (end of treatment).
Population: as for outcome 72
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 15 | 17 | 15
units on a scale
  Treatment Week 0 | 31.7 (9.7) | 32.8 (10.4) | 30.4 (10.1)
  Treatment Week 6 | 32.5 (13.0) | 29.6 (10.0) | 32.8 (10.9)
  Change | 0.8 (7.6) | -3.2 (4.6) | 2.4 (7.3)

77. Secondary Outcome: Neurocognitive Assessment Battery (MCCB) - Verbal Learning
Description: MCCB Verbal Learning domain score by week calculated from the Hopkins Verbal Learning Test-Revised, immediate recall (three learning trials only). The domain score scale is 20-80, with higher scores indicating a better outcome.
Time Frame: Once at Treatment Week 0 (baseline) and again at Treatment Week 6 (end of treatment).
Population: as for outcome 72
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 15 | 18 | 17
units on a scale
  Treatment Week 0 | 36.3 (8.5) | 33.4 (5.0) | 36.5 (8.2)
  Treatment Week 6 | 38.7 (9.9) | 35.8 (7.7) | 36.4 (4.4)
  Change | 2.5 (5.4) | 2.4 (5.8) | -0.1 (7.6)

78. Secondary Outcome: Neurocognitive Assessment Battery (MCCB) - Visual Learning
Description: MCCB Visual Learning domain score by week calculated from the Brief Visuospatial Memory Test-Revised. The domain score scale is 20-80, with higher scores indicating a better outcome.
Time Frame: Once at Treatment Week 0 (baseline) and again at Treatment Week 6 (end of treatment).
Population: as for outcome 72
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 15 | 18 | 17
units on a scale
  Treatment Week 0 | 33.8 (14.3) | 37.2 (10.8) | 35.1 (9.4)
  Treatment Week 6 | 36.2 (16.6) | 33.7 (10.0) | 34.2 (10.3)
  Change | 2.4 (6.2) | -3.4 (8.3) | -0.9 (7.2)

79. Secondary Outcome: Neurocognitive Assessment Battery (MCCB) - Working Memory
Description: MCCB Working Memory domain score by week calculated from the Wechsler Memory Scale, 3rd ed., spatial span subtest. The domain score scale is 20-80, with higher scores indicating a better outcome.
Time Frame: Once at Treatment Week 0 (baseline) and again at Treatment Week 6 (end of treatment).
Population: as for outcome 72
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 15 | 18 | 17
units on a scale
  Treatment Week 0 | 34.7 (10.7) | 33.7 (9.6) | 35.3 (11.0)
  Treatment Week 6 | 34.8 (11.1) | 34.7 (10.4) | 38.1 (11.7)
  Change | 0.1 (6.5) | 0.9 (7.7) | 2.8 (6.4)

80. Secondary Outcome: Positive and Negative Affect Schedule (PANAS) - Negative
Description: Participant reported responses after Brief Role Play rating how they felt during the role plays. Participants rated 12 negative affect items on a scale of 1-5, with 1 being "very slightly or not at all" and 5 being "extremely". The minimum score for this measure is 12 and the maximum score is 60. Higher scores indicate a higher rate of negative affect during the role plays.
Time Frame: Treatment Week 0 and Week 6
Population: Role play data was collected at baseline and week 6, so only those participants who completed the role play at week 6 appear in these outcome analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 15 | 17 | 17
units on a scale
  Treatment Week 0 | 20.5 (7.8) | 18.2 (7.0) | 20.2 (8.6)
  Treatment Week 6 | 18.8 (7.7) | 18.0 (5.6) | 18.9 (8.2)
  Change from Week 0 at Week 6 | -1.7 (5.7) | -0.2 (6.8) | -1.3 (5.6)

81. Secondary Outcome: Positive and Negative Affect Schedule (PANAS) - Positive
Description: Participant reported responses after Brief Role Play rating how they felt during the role plays. Participants rated 12 positive affect items on a scale of 1-5, with 1 being "very slightly or not at all" and 5 being "extremely". The minimum score for this measure is 12 and the maximum score is 60. Higher scores indicate a higher rate of positive affect during the role plays.
Time Frame: Treatment Week 0 and Week 6
Population: as for outcome 80
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 15 | 17 | 17
units on a scale
  Treatment Week 0 | 38.1 (8.6) | 37.0 (12.3) | 42.5 (8.9)
  Treatment Week 6 | 38.5 (12.8) | 39.5 (12.3) | 40.8 (9.6)
  Change from Week 0 at Week 6 | 0.4 (10.8) | 2.5 (11.4) | -1.6 (11.2)

82. Secondary Outcome: Reactions to Partner
Description: Participant reported responses after Brief Role Play. The Reactions to Partner item was calculated by totaling responses to 7 scales. Each scale score ranges from 1-5, which 1 being "completely agree" and 5 being "completely disagree". The minimum score for this measure is 7 and the maximum score is 35. Higher responses indicate a more negative reaction to their role play partner.
Time Frame: Treatment Week 0 and Week 6
Population: as for outcome 80
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 15 | 17 | 17
units on a scale
  Treatment Week 0 | 13.7 (4.2) | 14.4 (5.6) | 12.5 (4.2)
  Treatment Week 6 | 13.7 (3.1) | 13.9 (3.7) | 12.5 (3.5)
  Change from Week 0 at Week 6 | 0.0 (3.5) | -0.4 (4.0) | 0.0 (3.7)

83. Secondary Outcome: Willingness to Interact
Description: Participant reported responses after Brief Role Play. The Willingness to Interact item calculated by totaling scores from items 1-6. Each score ranges from 1-5, with 1 being "definitely willing" and 5 being "definitely unwilling". The minimum score for this measure is 6 and the maximum score is 30. Lower scores indicate more willingness to interact with their role play partner again in the future.
Time Frame: Treatment Week 0 and Week 6
Population: as for outcome 80
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Number analyzed (Participants) | 15 | 17 | 17
units on a scale
  Treatment Week 0 | 23.67 (4.13) | 23.18 (4.22) | 24.41 (4.33)
  Treatment Week 6 | 24.47 (3.31) | 24.24 (4.34) | 25.00 (4.29)
  Change from Week 0 at Week 6 | 0.80 (3.82) | 1.06 (3.60) | 0.59 (4.02)

ADVERSE EVENTS:
Arm/Group | 1: Oxytocin | 2: Galantamine | 3: Placebo
Serious Adverse Events (participants affected / at risk) | 0/17 | 1/20 | 0/21
Other Adverse Events (participants affected / at risk) | 4/17 | 1/20 | 0/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1: Oxytocin (N=17) | 2: Galantamine (N=20) | 3: Placebo (N=21)
hospitalization due to unrelated pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1: Oxytocin (N=17) | 2: Galantamine (N=20) | 3: Placebo (N=21)
Enuresis (Renal and urinary disorders) | 4 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No